CLINICAL TRIAL: NCT01276782
Title: Pilot Double-Blind Placebo Controlled Trial of Levothyroxine in Pregnant Systemic Lupus Erythematosus (SLE) Patients With Autoimmune Thyroid Disease
Brief Title: Levothyroxine in Pregnant SLE Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdraw the study because further analysis showed that it would be futile.
Sponsor: Johns Hopkins University (Other)
Collaborators: NYU Langone Health (Other); Duke University (Other); University of Chicago (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Michelle Petri M.D.,MPH, Professor of Medicine, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NA_00042993
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pregnant SLE (Placebo Comparator): Pregnant SLE patients with autoimmune thyroid antibodies will be randomized to levothyroxine or Placebo
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — It is FDA approved drug for thyroid disease

SUMMARY:
The last two decades have witnessed an explosion of new research documenting the deleterious impact that thyroid disease has on pregnancy and the postpartum period, in relation to miscarriage preterm delivery intelligence quotient of the unborn child and health of the mother postpartum. Both subclinical hypothyroidism and thyroid antibody positivity in euthyroid women have been associated with miscarriage and preterm delivery. Approximately 5% of all pregnant women have a thyroid disorder. both spontaneous miscarriage and preterm delivery.

Systemic lupus erythematosus (SLE), an autoimmune disorder of unknown etiology, has also been documented to negatively impact pregnancy. Women with Systemic lupus erythematosus (SLE)have increased rates of miscarriage and preterm delivery. Women with Systemic lupus erythematosus (SLE) also have increased rates of hypothyroidism and autoimmune thyroid disease (AITD, defined as the presence of thyroid antibodies with or without thyroid dysfunction). Preterm delivery (PTD), defined as birth prior to 37 weeks gestation, is the leading cause of neonatal mortality and morbidity in the United States. Although risk factors for preterm delivery exist, the majority of women have no known risk factors. Recently, both hypothyroidism and autoimmune thyroid disease have also been linked to preterm delivery. Given the increased prevalence of negative outcomes documented in pregnant women with thyroid disease, and the increased rates of hypothyroidism and Autoimmune thyroid disease in women with Systemic lupus erythematosus (SLE), the investigators determined that Autoimmune thyroid disease was associated with both preterm delivery and miscarriage. This has led to this application to begin a pilot randomized clinical trial of thyroxine in autoimmune thyroid disease in systemic lupus erythematosus pregnancy.

DETAILED DESCRIPTION:
Objectives: The investigators hypothesize that levothyroxine decreases miscarriages and preterm birth.

The investigators will compare levothyroxine versus placebo to determine the effects on pregnant women with Autoimmune thyroid disease.

Background:The last two decades have witnessed an explosion of new research documenting the deleterious impact that thyroid disease has on pregnancy and the postpartum period, in relation to miscarriage, preterm delivery , Intelligence quotient (IQ) of the unborn child and health of the mother postpartum . Both subclinical hypothyroidism and thyroid antibody positivity in euthyroid women have been associated with miscarriage and preterm delivery. .Even minor perturbations of thyroid function have been linked to decreased Intelligence Quotients and impaired neurological development of the unborn child. Approximately 5% of all pregnant women have a thyroid disorder (either subclinical or overt hypothyroidism or hyperthyroidism). Intervention in pregnancy with levothyroxine in euthyroid thyroid antibody positive women has been shown in a prospective study, performed in an area of mild iodine deficiency, to significantly decrease the rate of both spontaneous miscarriage and preterm delivery .

SLE has also been documented to negatively impact pregnancy. Women with systemic lupus erythematosus (SLE) have increased rates of miscarriage and preterm delivery, especially in the setting of active Systemic lupus erythematosus and antiphospholipid antibodies . The offspring of women with Systemic lupus erythematosus are at increased risk for heart block and require neonatal intensive care unit care more frequently . Furthermore, pregnant women with Systemic lupus erythematosus (SLE) have increased mortality rates. Women with Systemic lupus erythematosus (SLE) also have increased rates of hypothyroidism and autoimmune thyroid disease (AITD, defined as the presence of thyroid antibodies with or without thyroid dysfunction). In a recent case-control study performed by questionnaire, Yuen et al documented a 21% prevalence of thyroid disease in Systemic lupus erythematosus (SLE) women versus 10% in controls (p=0.02).

Preterm delivery (PTD), defined as birth prior to 37 weeks gestation, is the leading cause of neonatal mortality and morbidity in the United States. Despite a public health effort to decrease the prevalence of Preterm Delivery (PTD) , the prevalence has increased from 11% in 1996 to 12.7% in 2007, with an annual societal cost of over 26 billion dollars. In an attempt to affect the societal impact of preterm delivery, the Surgeon General made decreasing the prevalence of Preterm Delivery to 7.6% a goal of Healthy People 2010. Although risk factors for Preterm Delivery exist, the majority of women have no known risk factors. Recently, both hypothyroidism and autoimmune thyroid disease have also been linked to preterm delivery.

Given the increased prevalence of negative outcomes documented in pregnant women with thyroid disease, and the increased rates of hypothyroidism and Autoimmune thyroid disease in women with systemic lupus erythematosus, the investigators previously evaluated the prevalence of thyroid disease during pregnancy and postpartum in women with systemic lupus erythematosus, as well as pregnancy outcome. The investigators determined that autoimmune thyroid disease was associated with both preterm delivery and miscarriage in the Hopkins Lupus Cohort . This has led to this application to begin a pilot randomized clinical trial of levothyroxine in autoimmune thyroid disease in Systemic Lupus Erythematosus pregnancy.

Preliminary Data:

The prevalence of thyroid antibody positivity was 31.5%. Preterm birth was strongly associated with Autoimmune Thyroid Disease in systemic lupus erythematosus (p=0.002). The investigators found: 1) a high percentage of women (13%) were on thyroid hormone replacement prior to becoming pregnant, 2) a high percentage of women (10.9%) presented with previously undiagnosed subclinical hypothyroidism during pregnancy, 3) 14% of women developed postpartum thyroiditis, 4) antibody positivity during pregnancy was not predictive of the occurrence of postpartum thyroiditis, and 5) women with thyroid disease had a dramatic increase in the prevalence of preterm delivery as compared to women who had no thyroid disease. Overall, the percentage of women with systemic lupus erythematosus who either had levothyroxine treated thyroid disease prior to pregnancy, who were diagnosed with thyroid disease during pregnancy, or who developed postpartum thyroiditis, was 37.9%. None of the demographic, laboratory, medication usage, or disease activity index data affected the association of autoimmune thyroid disease with adverse pregnancy outcome.

Significance:

Preterm delivery was markedly increased in the group of Systemic Lupus Erythematosus women who had thyroid disease diagnosed either prior to, during, or in the postpartum period, as compared to the group of women who were thyroid disease free, in our previous study. Our results were not affected by the dosage of prednisone administered or the cardiolipin antibody titer. Furthermore, the increased rate of preterm delivery in the Systemic Lupus Erythematosus women with thyroid disease was not secondary to Systemic Lupus Erythematosus activity, as the Physician Global Assessment score and Systemic Lupus Erythematosus Disease Activity Index were similar in Systemic Lupus Erythematosus women with or without thyroid disease. These results are consistent with a growing body of evidence linking thyroid disorders, both hypothyroidism and autoimmune thyroid antibodies in euthyroid women, to Preterm delivery .

In conclusion, women with Systemic Lupus Erythematosus have a high prevalence of primary hypothyroidism,undiagnosed subclinical hypothyroidism, and postpartum thyroiditis. In sum, a minimum of one in every three pregnant women with systemic lupus erythematosus falls into one of these categories. Autoimmune thyroid disease is highly associated with adverse pregnancy outcomes.

Our current application will begin a pilot trial of levothyroxine versus placebo at the United States sites with a long track record of interest in Systemic Lupus Erythematosus and pregnancy.

Study Procedures Systemic lupus erythematosus (SLE) will be defined by the American College of Rheumatology (ACR) classification criteria or by the Systemic Lupus International Collaborative Clinics revised American College of Rheumatology criteria. Systemic lupus erythematosus (SLE) patients already on levothyroxine and those discovered to be hypothyroid needing levothyroxine, will be excluded.

Pregnant Systemic lupus erythematosus patients with autoimmune thyroid antibodies who give informed consent will be randomized to levothyroxine (50mcg) versus placebo.

Outcome measures will follow those used in the Predictors of Pregnancy Outcome: Biomarkers in Anti-Phospholipid Antibody Syndrome (APS) and Systemic Lupus Erythematosus (SLE) (PROMISSE) study. The outcome will be adverse pregnancy outcome (preterm birth, miscarriage, or stillbirth).

The endpoint is adverse pregnancy outcome as defined by the Promisse study

The composite endpoint defined as the occurrence of one or more of the following events:

1. Otherwise unexplained fetal death occurring after 12 weeks gestation
2. Neonatal death prior to hospital discharge and due to complications of prematurity
3. Indicated preterm delivery prior to 36 weeks' gestation because of gestational hypertension, preeclampsia-eclampsia, or placental insufficiency
4. Intrauterine growth restriction (IUGR) Enrollment will be at Johns Hopkins Hospital, Hospital for Joint Diseases (Jill Buyon M.D.) Oklahoma Medical Research Foundation (Joan Merrill M.D.), University of Chicago (Tammy Utset M.D., M.P.H.) Duke University Medical Center (Megan Clowse M.D., M.P.H) and Stanford University (Eliza F. Chakravarty, M.D.). Dr D. Ware Branch at the University of Utah will be the gynecologic consultant to adjudicate the outcomes.

TSH testing will be performed using the Ultrasensitive hTSH II method on an AbbottAxsym. (Abbott Diagnostics, Abbott Park, Illinois.) This is a Microparticle Enzyme Immunoassay (MEIA) method. The analytical sensitivity of the Axsym Ultrasensitive hTSH II is 0.03 uIU/mL. The intraassay coefficient of variation (CV) is 4.35% and the interassay coefficient of variation (CV) is 5.73%. A TSH greater than 2.5 μU/ml in the first trimester, or greater than 3.0 μU/ml in the second or third trimester was considered abnormal. Glinoer et al has demonstrated that 18% of women without thyroid disease have a suppressed Thyroid Stimulating Hormone (TSH) . Therefore, in our previous study TSH values below 0.3 μU/ml were not considered abnormal during pregnancy unless it occurred after the 20th week of gestation.

Serum thyroglobulin antibody (Tg-Ab) and thyroid peroxidase antibody (TPO-Ab) , also research test, will be measured by enzyme-linked immunosorbent assay (KRONUS KalibreTM Thyroglobulin Antibody and Thyroid Peroxidase Antibody ELISA kits will be kindly provided by KRONUS Corp, Boise, ID). Serum anti-Tg levels above 3 U/mL were considered positive and anti-TPO levels above 2 U/mL will be considered positive.

Study duration and number of study visits required of research participants:

The study duration is upto 36 weeks of pregnancy after screening. The patient will be seen monthly using the accepted clinical guidelines devised for the PROMISSE (Predictors of Pregnancy Outcome: Biomarkers in Anti-Phospholipid Antibody Syndrome (APS) and Systemic Lupus Erythematosus (SLE)) study, an National Institute of Health funded prospective study of the role of the antiphospholipid antibodies in pregnancy. At each pregnancy visit, the Stemic Lupus Erythematosus Pregnancy Disease Activity Index (SLEPDAI), physician global assessment, blood pressure, urine protein to creatinine ratio,Complement 3 (C3) ,Complement 4 (C4) and anti-double stranded DNA will be recorded. Anticardiolipin and lupus anticoagulant will be recorded as part of standard of care. All women will be followed by both their rheumatologist and their obstetrician.

Plan for reporting unanticipated problems or study deviations. The Data Safety Monitoring Committee will review all adverse events monthly. All serious adverse events will be reported per Federal and JHM-IRB regulations Definition of treatment failure or participant removal criteria. Treatment failure does not apply.

1. Systemic lupus erythematosus (SLE) patients who experience an allergic reaction to Levolevothyroxine.
2. Patients who fail to adhere to study instructions.
3. Patients who develop medium to severe adverse events.
4. Withdrawal of consent.
5. A patient with clinical hypothyroidism, elevated Thyroid Stimulating Hormone or clinical hyperthyroidism

5. Inclusion/Exclusion Criteria Inclusion Criteria All Systemic lupus erythematosus (SLE) pregnant women (aged 18 - 45 years) before 14 weeks of gestation, with autoimmune thyroid antibodies Exclusion Criteria

* Systemic lupus erythematosus (SLE) patients already on levothyroxine.
* Those patients discovered to be hypothyroid who need levothyroxine as part of standard of care 6. Drugs/ Substances/ Devices In a prospective study Negro et. al has demonstrated that thyroxin given to women with antithyroid antibodies significantly decreased the rate of both spontaneous miscarriage and preterm. The investigators plan to administer the drug/placebo only for the duration of the pregnancy.

The dose will be 50 mcg daily.

ELIGIBILITY:
Inclusion Criteria:

* All SLE (Systemic Lupus Erythematosus) pregnant women (aged 18 - 45 years) before 14 weeks of gestation, with autoimmune thyroid antibodies

Exclusion Criteria:

* SLE (Systemic Lupus Erythematosus) patients already on levothyroxine. Those patients discovered to be hypothyroid who need levothyroxine as part of standard of care

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
preterm birth | Delivery prior to 36 weeks

SECONDARY OUTCOMES:
Miscarriage | Loss of fetus before 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Petri, MD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States